CLINICAL TRIAL: NCT00465166
Title: Lumbar Spine Ultrasound of Patients With Previous Accidental Dural Puncture During Labour Epidural
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Other Study IDs: 07-05; 07-0002-E
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Postdural Puncture Headache
Keywords: Accidental dural puncture; Labour epidural; Ultrasound; Ligamentum flavum
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who had a documented, accidental dural puncture during placement of their labor epidural.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Lumbar ultrasound from L1-S1, carried out using a portable ultrasound system equipped with a 2-5 MHz curved array probe.

SUMMARY:
Accidental dural puncture is a potential complication of epidural analgesia for labour and delivery. When it happens, it may cause debilitating headaches and other symptoms that prevent mothers from talking care of their newborns. Accidental dural puncture is related to the operator performance and to individual anatomical variations of the spine. The purpose of this study is to do a lumbar spine ultrasound on the patients who have had accidental dural punctures and analyze if there is any abnormal anatomy seen. Then, we will compare the position of any spinal abnormality to the position of the dural puncture reported in the anaesthesia record.

DETAILED DESCRIPTION:
Effective epidural analgesia depends on accurate identification of the epidural space for delivery of analgesic mixtures. The technique of loss of resistance to either saline or air is the most commonly used method to locate the epidural space. Although this technique has a high success rate, it is associated with a significant incidence of accidental dural punctures. Accidental dural punctures might be related to the operator performance or to individual anatomical variations.

A normal ligamentum flavum is fundamental in the loss of resistance technique. However, many cadaver dissection and radiological studies in the literature have showed that the ligamentum flavum may in fact not fuse at the midline; thereby leaving a gap between its left and right portions. Ligamentum flavum midline gaps are thought to be a potential cause of failed recognition of loss of resistance during epidural needle placement and consequently accidental dural puncture. Therefore, if it were feasible to avoid inserting the epidural needle at the same level where a ligamentum flavum midline gap exists, then dural punctures may be less likely.

Lumbar spine ultrasound has been very useful in consistently identifying important anatomical landmarks for epidural needle placement including the ligamentum flavum. It is unknown at this time whether ultrasound is a useful modality to detect abnormal anatomy. Our study will evaluate by ultrasound scan the lumbar vertebral column of patients who have had a previously recognized accidental dural puncture. Our objective is to determine whether or not there is a correlation between accidental dural punctures and abnormalities of ligamentum flavum as seen by ultrasound imaging. Our hypothesis is that patients who have had accidental dural punctures have abnormal anatomy of ligamentum flavum that can be detected by lumbar spine ultrasound.

Lumbar ultrasound imaging from L1-S1 will be performed with the patient in the sitting position. The best possible image captured at the transverse approach for each of the interspaces from L5-S1 to L1-L2 will be saved for analysis of both ligamentum flavum (primary outcome) and symmetry (secondary outcome). A normal ligamentum flavum is described as a hyperechoic continuous midline band, which is aligned with the hyperechoic signal of the transverse processes. An abnormal ligamentum flavum will be described as a non-continuous or even absent signal. The presence of symmetric anatomy is defined as an equal distant between the left and right articular processes and the transverse processes to the midline.

Incidence of abnormal ligamentum flavum and asymmetry will be presented in a descriptive way and the level of anatomical abnormality detected by ultrasound will be correlated to the level of dural puncture reported on the anaesthesia record.

ELIGIBILITY:
Inclusion Criteria:

* Previous dural puncture during labour epidural

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had a documented, accidental dural puncture during placement of their labor epidural.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2007-02; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada